CLINICAL TRIAL: NCT00163124
Title: A Randomized Controlled Trial of Best Approach to Care Compared to Diversified Adjustive Technique
Brief Title: A Randomized Controlled Trial of Best Approach to Care Compared to Diversified Chiropractic Adjustive Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker College of Chiropractic (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PCC2005-003
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Low Back Pain; Headache; Shoulder Pain
Keywords: chiropractic; spinal manipulation; low back pain
MeSH Terms: conditions — Low Back Pain; Headache; Shoulder Pain | interventions — Manipulation, Spinal; Patient Education as Topic; Nutritional Status

INTERVENTIONS:
Procedure: spinal manipulation & patient education/nutrition

SUMMARY:
There are a variety of treatment approaches used by the chiropractic profession. Some of these require forceful joint manipulation and some do not. This study is designed to compare outcomes of two such techniques that are common to chiropractic practice. The hypothesis is that there is no difference between forceful and non-forceful approaches to treatment.

DETAILED DESCRIPTION:
The comparison will permit a one month treatment period for both techniques and a three week follow-up. Patients will be assessed at baseline (intake), and at specified intervals and at three weeks following the termination of care.

ELIGIBILITY:
Inclusion Criteria:

chronic musculoskeletal pain ability to communicate in English

Exclusion Criteria:

pregnancy contraindications to manipulation pending litigation chiropractic care within the last month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155
Dates: Start 2005-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Pain Disability Index (PDI)

SECONDARY OUTCOMES:
Beck Depression Inventory
Patient Expectation
Evaluation of Clinic Services

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hawk, PhD DC, Principal Investigator — Parker College of Chiropractic
Locations (1):
- Parker College of Chiropractic, Dallas, Texas, United States